CLINICAL TRIAL: NCT00738192
Title: Comparison of Analgesic Efficacy of Fentanyl, Sufentanil and Butorphanol After Remifentanil Anesthesia in Gynecological Laparoscopic Surgeries
Brief Title: Comparison of Analgesic Efficacy of Fentanyl, Sufentanil and Butorphanol After Remifentanil Anesthesia
Acronym: CARAN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Responsible Party: XiaoFeng Shen, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NMU-FY2008-311; NJFY0807311M
Record Dates: First submitted 2008-08-18; First posted 2008-08-20 (Estimated); Last update posted 2009-03-11 (Estimated); Status verified 2009-03

CONDITIONS: Postoperative Pain
Keywords: Postoperative analgesia; Opioids; Laparoscopic surgery
MeSH Terms: conditions — Pain, Postoperative | interventions — Fentanyl; Sufentanil; Butorphanol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Fentanyl delivered for controlling awaking pain
  Interventions: Drug: Fentanyl citrate
- 2 (Active Comparator): Sufentanil delivered for controlling awaking pain
  Interventions: Drug: Sufentanil citrate
- 3 (Active Comparator): Butorphanol delivered for controlling awaking pain
  Interventions: Drug: Butorphanol tartrate

INTERVENTIONS:
Drug: Fentanyl citrate — Fentanyl 0.5 μg/kg delivered intravenously immediate at the end of remifentanil pump finished
  Other Names: Fentanil
  Arms: 1
Drug: Sufentanil citrate — Sufentanil 0.05 μg/kg delivered intravenously immediate at the end of remifentanil pump finished
  Other Names: Sufenil
  Arms: 2
Drug: Butorphanol tartrate — Butorphanol 0.01 mg/kg delivered intravenously immediate at the end of remifentanil pump finished
  Other Names: Nuoyung
  Arms: 3

SUMMARY:
Fast awakening from anesthesia is one of the major characteristics of remifentanil-associated anesthetic induction and maintenance, whereas corresponding pain during awakening influences patient's rehabilitation strongly. In addition, such early postoperative pain results in significant stress responses, which displays as further release of stress hormones such as cortisol and β-endorphin as well. How to prevent such acute pain resulting from remifentanil's fast metabolism endows clinical significance. This study is designed to compare the analgesic efficacy of fentanyl, sufentanil and butorphanol delivered after gynecological laparoscopic surgeries that underwent remifentanil induction and maintenance, and investigate corresponding influence on the levels of blood cortisol and β-endorphin.

ELIGIBILITY:
Inclusion Criteria:

1. ASA physical status I-II
2. Chinese
3. 19-45yr
4. Selective laparoscopic surgeries

Exclusion Criteria:

1. Allergy to opioids, a history of the use of centrally-acting drugs of any sort, chronic pain and psychiatric diseases records
2. Participants younger than 18 years, older than 45 years or pregnancy was eliminated
3. Due to the significant changes in vital signs might affect cognition of pain and that of sensation, over 20% variation of these records from the baselines or below 92% of SpO2 under 20-40% nasal tube oxygen at any time should be excluded from the study
4. Those who were not willing to or could not finish the whole study at any time

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2008-07; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
VAS ratings of pain | 0 min after awake from anesthesia; 5,10,15,20 and 30min after awake from anesthesia

SECONDARY OUTCOMES:
Hemodynamics of patients | 30min before operation; every 10min during operation; 5,10,15,20,30 and 60min after operation
Sedative ratings with VAS system | 0,5,10,15,25,45 and 60min after awake from anesthesia
Overall VAS satisfaction ratings | 1 h after operation
Blood cortisol and β-endorphin levels | 0, 10min before the end of surgeries, 10min, 1h and 6h after operation
Side effects | 1 h after operation

CONTACTS AND LOCATIONS:
Overall Officials: XiaoFeng Shen, MD, Study Chair — Nanjing Medical University
Locations (1):
- Nanjing Maternal and Child Health Care Hospital, Nanjing, Jiangsu, China